CLINICAL TRIAL: NCT05888116
Title: Clinical Investigation to Evaluate the Efficacy and Safety of a Hyaluronic Acid-Based Vaginal Moisturizer Medical Device to Ease Symptoms of Vaginal Dryness
Brief Title: Efficacy and Safety of a Hyaluronic Acid-Based Vaginal Moisturizer Medical Device to Ease Symptoms of Vaginal Dryness
Acronym: HYALU-LAUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dermofarm, S.A.U (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFARM-HYDRA-HA-2022
Record Dates: First submitted 2023-05-09; First posted 2023-06-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-09

CONDITIONS: Vaginal Disease
Keywords: Vaginal Disease; Vaginal Dryness; Vaginal Atrophy
MeSH Terms: conditions — Vaginal Diseases

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, controlled, double-blind study with two parallel group of subjects. The clinical investigation will be performed in 9 clinical sites.
  The follow-up will be 4 weeks, with 3 face-to-face controls (baseline, 7 days and 30 days) and 2 telephone controls (3 days and 21 days).
  At all on-site visits (baseline, Day 7, Day 30), the investigator will record the severity of patient-reported symptoms (via VAS of 0 to 100 mm) and perform a gynecological examination to evaluate signs of vaginal atrophy. Potential adverse events and potential device deficiencies will be recorded at each visit.
  The patients will have a patient notebook where they will record the intensity of the symptoms on the third day and weekly, as well as the possible appearance of adverse events or product deficiencies.
Who Masked: Participant, Investigator
Masking Description: To maintain the double-blind, both the investigational and comparator products will be dispensed in white boxes, labeled with the study code and the patient code. Each patient code will be assigned to one treatment or the other according to a predetermined randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hidratante HA (Experimental): The investigational product consists of a new vaginal moisturizing gel (class IIb medical device) presented in the form of 5 ml single-dose containers. Each patient will be given 12 single-dose containers inside white boxes identified only with the patient code.
  For each participant, the total duration of treatment will be 4 weeks.
  Interventions: Device: Hidrante HA
- Cumlaude Hidratante Interno® (Active Comparator): The investigational product is a marketed vaginal moisturizing gel (class IIb medical device) presented in the form of 5 ml single-dose containers. Each patient will be given 12 single-dose containers inside white boxes identified only with the patient code.
  For each participant, the total duration of treatment will be 4 weeks.
  Interventions: Device: Cumlaude Hidrante Interno®

INTERVENTIONS:
Device: Hidrante HA — Apply the 5 ml single dose three times a week, every other day, preferably at night before going to bed for 4 weeks.
  Other Names: Experimental
  Arms: Hidratante HA
Device: Cumlaude Hidrante Interno® — Apply the 5 ml single dose three times a week, every other day, preferably at night before going to bed for 4 weeks.
  Other Names: Active comparator
  Arms: Cumlaude Hidratante Interno®

SUMMARY:
This study evaluates the efficacy and safety of a new hyaluronic acid-based vaginal moisturizer gel to ease symptoms of vaginal dryness compared to a commonly used marketed vaginal moisturizer (Cumluade Hidratante Interno®).

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, controlled, double-blind clinical investigation to evaluate the safety and efficacy of a new hyaluronic acid-based vaginal moisturizer gel (medical device class IIb) in women with symptoms of vaginal atrophy and dryness, compared to a commonly used marketed vaginal moisturizer in gynecology clinics (Cumluade Hidratante Interno®), with a 1-month follow-up.

The participants will apply the single dose of vaginal moisturizer 3 times per week, every other day, preferably in the evening.

The investigators will monitor the evolution of vaginal symptoms, vaginal health using the Vaginal Health Index (VHI), sexual function using the Female Sexual Function Index (FSFI) questionnaire, and the safety and tolerability of the new class IIb medical device.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age who manifest subjective symptoms of vaginal dryness (dryness, itching, burning/stinging and dyspareunia).
* In the case of postmenopausal women, they must have a diagnosis confirmed by the gynecologist of the presence of signs of vulvovaginal dryness/atrophy (Vaginal Health Index score <15).
* Patients who have not used any topical treatment, moisturizer or vaginal lubricant for at least 7 days prior to the start of the study and agree not to use it during the study period.
* Patients who agree to participate and sign the Informed Consent form.

Exclusion Criteria:

* Pregnant women
* Malignant neoplasm within 5 years prior to study entry (except for treated basal cell/squamous cell carcinoma of the skin).
* Genital bleeding.
* Treatment with vaginal or systemic estrogens in the 3 months prior to study inclusion or during the study period. I said above
* Subjects with illness or other medical condition that, in the investigator's opinion, would compromise participation or could lead to hospitalization during the study.
* Clinical evidence of acute infection that requires treatment (syphilis, herpes simplex, human papilloma virus, gonorrhea, chlamydia, lymphogranuloma venereum, etc.); clinical evidence or history of chronic infectious disease (i.e., tuberculosis), with the exception of HPV-carrying women with no lesions.
* Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt or suicidal ideation, or any other psychiatric illness (except intermittent anxiety).
* Known allergy to the components of the investigational product or its excipients.
* Drug or alcohol abuse in the 12 months prior to the start of the study.
* Participation in an interventional clinical study or administration of any investigational agent within the previous 30 days.
* Patients with low expectation of compliance with the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female can have vaginal disease.
Enrollment: 54 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Vaginal Health Index | At the end of study (Day 30)
  The Vaginal Health Index ranges from a minimum of 5 to a maximum of 25. The change will be assessed by comparing scores from baseline to 30 days (final visit); with comparison intra and inter groups.

SECONDARY OUTCOMES:
Severity of subjective symptoms (investigator record) | at 7 days and 30 days.
  Severity of dryness, itching, burning and dyspareunia reported by the investigator in the data registration form, assessed using a visual analog scale (VAS from 0=none to 10=maximum).The change will be assessed by comparing scores from baseline to day 7 and to day 30; with comparison intra and inter groups.
Subjective symtomps (patient's notebook) | at 3 days, 7days, 14 days, 21 days and 30 days.
  Severity of dryness, itching, burning and dyspareunia reported on patient diary using a 4-point Likert scales (0 = absent, 1 = mild, 2 = moderate, and 3 = severe). The change will be assessed by comparing scores from baseline to every record (3 days, 7days, 14 days, 21 days and 30 days); with comparison intra and inter groups.
Objective signs of vulvovaginal atrophy | at 7 days and 30 days.
  Objective signs of vulvovaginal atrophy (dryness, flattening of folds, mucosal pallor, frailty and petechiae) reported by the investigator in the data registration form, assessed using a 4-point Likert scales (0 = absent, 1 = mild, 2 = moderate, and 3 = severe). The change will be assessed by comparing scores from baseline to day 7 and to day 30; with comparison intra and inter groups.
Vaginal pH | At the end of study (Day 30)
  Vaginal pH will be measured by the investigator with a test strip delivered by sponsor. The change will be assessed by comparing pH values from baseline to day 30; with comparison intra and inter groups.
Sexual function | At the end of study (Day 30)
  Female Sexual Function Index (FSFI) questionnaire will be answered by the patients at the baseline and 30-day visits. The change will be assessed by comparing FSFI scores from baseline to day 30; with comparison intra and inter groups.
Global Symptom Score (GSS) | At the end of study (Day 30)
  Global Symptom Score (GSS) will be assessed by the sum of severity scores of each symptom: dryness, itching, burning/stinging and dyspareunia (0 = none, 1 = mild, 2 = moderate and 3 = severe). GSS score ranges from 0 to 12. The change will be assessed by comparing GSS scores from baseline to day 30; with comparison intra and inter groups.
Adverse events as a measure of Safety and Tolerability | At the end of study (Day 30)
  Number of participants with incidence of treatment-related adverse events, serious adverse events and device deficiencies as a Measure of Safety and Tolerability.
Overall Safety Assessment | At the end of study (Day 30)
  Overall patient and investigator safety rating, using 4-point Likert-type scale (1 = very good, 2 = good, 3 = moderate, 4 = poor, 5=very poor); with comparison inter groups.
Patient satisfaction | At the end of study (Day 30)
  The patient's degree of satisfaction with the product will be rated using a 5-point Likert-type scale (1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5=very dissatisfied); with comparison inter groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fasero, Ph, Principal Investigator — Clínica Corofas. Tomelloso. Ciudad Real
Locations (1):
- Corofas Menopause, Tomelloso, Ciudad Real, Spain